CLINICAL TRIAL: NCT00006337
Title: Adenosine A2A Blockade With KW-6002 in Parkinson's Disease
Brief Title: KW-6002 to Treat Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010001; 01-N-0001
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Parkinson's Disease
Keywords: Clinical Trial; Dyskinesias; Levodopa Infusion
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — istradefylline; Levodopa

INTERVENTIONS:
Drug: KW-6002
Drug: IV Levodopa

SUMMARY:
This study will evaluate the effects of an experimental drug called KW-6002 on Parkinson's disease symptoms and on dyskinesias (involuntary movements) that develop as a result of long-term treatment with levodopa. This drug blocks the action of the neurotransmitter adenosine, thought to be involved in producing Parkinson's symptoms.

Patients with relatively advanced (Stage II to IV) Parkinson's disease between 30 and 80 years of age may be eligible for this 7-week study. Participants will have a complete medical history and physical examination, including blood tests and an electrocardiogram, and possibly brain magnetic resonance imaging (MRI), CT scan, and chest X-ray.

Patients enrolled in the study will, if possible, stop taking all antiparkinsonian medications except levodopa (Sinemet) for one month before the study begins and throughout its duration. For the first 1 to 3 days, patients will be admitted to the NIH Clinical center to undergo a levodopa "dose-finding" procedure. For this study, patients will stop taking Sinemet and instead will have levodopa infused through a vein for up to 8 hours/day. During the infusions, the drug dose will be increased slowly until either 1) parkinsonian symptoms improve, 2) unacceptable side effects occur, or 3) the maximum study dose is reached. Symptoms will be monitored frequently to find two infusion rates: 1) one that is less than what is needed to relieve symptoms, and 2) one that relieves symptoms but may produce dyskinesias. This procedure will be repeated at the end of weeks 2, 4 and 6 of the study.

When the patient's optimal dose is determined treatment will begin. Patients will take tablets or capsules containing KW-6002 or placebo (a look-alike pill with no active ingredient) once a day for 2 weeks, in addition to their regular Sinemet. All participants will receive placebo at least 2 weeks during the study; some patients will receive only placebo throughout the entire 7 weeks. At the end of weeks 1, 3 and 5, patients will be evaluated with a brief physical examination, routine blood and urine tests, and assessment of any adverse effects.

Throughout the study, parkinsonian symptoms and dyskinesias will be evaluated and blood samples will be drawn periodically to measure drug levels.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the acute effects of adenosine A2a receptor blockade on parkinsonian symptoms and levodopa-associated motor response complications in patients with advanced Parkinson's disease. In a controlled clinical trial, efficacy will be assessed through the use of validated motor function scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
Males and females between the ages of 30-80.

Carry the diagnosis of idiopathic Parkinson's disease based on the presence of a characteristic clinical history and neurologic findings.

Patients with relatively advanced disease (Hohen and Yahr stage II-IV in the off state).

Patients with Parkinson's disease who have been treated with levodopa for at least one year.

Patients with Parkinson's disease who require levodopa/carbidopa dosing at qid or more frequent intervals.

Will have been receiving a stable regimen of treatment for Parkinson's disease for at least 4 weeks prior to study admission.

Patients with Parkinson's disease who have associated motor response complications, including wearing-off fluctuations and peak-dose dyskinesias.

Must be able to provide written informed consent.

Patients with non-idiopathic parkinsonism or parkinsonian variants (e.g. juvenile Parkinson's disease; atypical parkinsonism; secondary parkinsonism; progressive supra-nuclear palsy; Shy-Drager syndrome; olivopontocerebellar atrophy will be excluded.

Patients with a clinically significant illness of any organ system, including hepatic, renal, pancreatic, cardiovascular, endrocrinologic, gastrointestinal, respiratory, and neurologic system (except for those with Parkinson's disease) who may require a change in the treatment of that illness during the trial, or that may compromise the safety of the patient volunteer during the trial, or that may affect the ability of the volunteer to complete the trial will be excluded.

No presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk, including cancer (except basal cell carcinoma or surgically excised carcinoma in situ of the cervix) as well as liver or pancreatic enzyme test results above the upper limit of normal.

Patients who have had bilateral intracranial neurosurgical procedures such as nuclear ablation, stimulator implantation or tissue transplantation will be excluded.

Patients with a history of seizures, including one or more infantile febrile seizures, or with a history of neuroepileptic malignant syndrome will be excluded.

Patients who, for any reason, are judged by the investigator to be inappropriate for the study (including volunteers who are unable to communicate or to cooperate with the investigator) will be excluded.

Patients with significant dementia (MMSE 25 or less), major psychotic illness, history of drug or alcohol abuse within past two years, and those who require drug therapy for a DSM-IV major depressive episode will be excluded.

Patients who satisfy DSM-IV criteria for alcohol or other drug abuse or dependence within two years of being exposed to KW-6002 will be excluded.

Patients who have been treated with a centrally acting dopamine antagonist drug, including neuroleptic agents, metoclopramide and buspirone within three months (within six months for depot formulations) because of the potential liability for extrapyramidal side effects will be excluded.

Patients taking nonselective monoamine oxidase inhibitors (phenelzine, isocarboxazid, tranylcypromine) will be excluded.

Patients who have taken terfenadine, astemizole, cisapride, simvastatin, lovastatin, felodipine, or nifedipine within seven days before being exposed to KW-6002 will be excluded.

Patients who have previously been exposed to KW-6002 or who have been treated with any other investigational agents within 12 weeks (or within five half-lives for investigational agents with a half-life of longer than 2 weeks) of being exposed to KW-6002 will be excluded.

Patients with unacceptable prior/concomitant medications as will patients who have taken an investigational drug within the 2 months prior to randomization will be excluded.

Pregnant will be excluded.

Females who are of childbearing potential must be using a reliable method of contraception at the time they agree to study participation and must agree to continue using a reliable method of contraception include hormonal products (e.g. approved oral contraceptives or long-term injectable or implantable contraceptives), double barrier methods (e.g. condom plus diaphragm; condom plus spermicidal foam; condom plus spermicidal sponge). an intra-uterine device or tubal ligation.

All female volunteers of child-bearing potential must have a negative urine pregnancy test on the day before first exposure to KW-6002.

No patients taking any medications listed in Section 6.2, Forbidden Medications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 2000-10; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Chase TN, Oh JD, Blanchet PJ. Neostriatal mechanisms in Parkinson's disease. Neurology. 1998 Aug;51(2 Suppl 2):S30-5. doi: 10.1212/wnl.51.2_suppl_2.s30. PMID 9711978
- [Background] Mizuno Y, Mori H, Kondo T. Parkinson's disease: from etiology to treatment. Intern Med. 1995 Nov;34(11):1045-54. doi: 10.2169/internalmedicine.34.1045. PMID 8774962
- [Background] Bernheimer H, Birkmayer W, Hornykiewicz O, Jellinger K, Seitelberger F. Brain dopamine and the syndromes of Parkinson and Huntington. Clinical, morphological and neurochemical correlations. J Neurol Sci. 1973 Dec;20(4):415-55. doi: 10.1016/0022-510x(73)90175-5. No abstract available. PMID 4272516